CLINICAL TRIAL: NCT02455739
Title: Effect of Gum Chewing on Intestinal Functions After Gynecologic Operations
Brief Title: Gum Chewing and Postoperative Intestinal Function After Gynecolgic Operations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, enis ozkaya, medical doctor, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZEYNEP KAMIL
Record Dates: First submitted 2015-05-20; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Gastrointestinal Disorder Postoperative
Keywords: intestinal function; chewing gum
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chewing gum positive (Experimental): chewing gum group will chew gum
  Interventions: Other: chewing gum
- chewing gum negative (No Intervention): chewing gum group will not chew gum

INTERVENTIONS:
Other: chewing gum — postoperative gum chewing to improve gastrointestinal function
  Arms: chewing gum positive

SUMMARY:
The investigators aimed to assess whether postoperative gum chewing improve intestinal functions.

DETAILED DESCRIPTION:
We will randomize patients into two groups after gynecologic operations. One group will chew gum, the other group not and we will assess the gastrointestinal function functions.

ELIGIBILITY:
Inclusion Criteria:

* Women underwent gynecologic operation
* Women who are eligible for gum chewing

Exclusion Criteria:

* Women with previous gastrointestinal intervantion
* Women with previous abdominal surgery

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Gastrointesitinal function | postoperative first 48 hours
  Gastrointesitinal function will be assess by bowel sound for every 2 hours and time of flatulence will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Ateş Karateke, md, Study Director — Zeynep Kamil
Locations (1):
- Zeynep Kamil, Istanbul, Turkey (Türkiye)